CLINICAL TRIAL: NCT03163745
Title: Asymptomatic Spontaneous Bacterial Peritonitis in Patients With Decompensated Liver Cirrhosis in Upper Egypt : A Prospective Hospital Based Study
Brief Title: Asymptomatic Spontaneous Bacterial Peritonitis in Patients With Decompensated Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Antony Albair Georgy, AssiutU, Assiut University
Other Study IDs: ASBP
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Paracentesis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic spontaneous bacterial peritonitis: All the included patients will be subjected to:
  1. Full medical History and physical examination
  2. Laboratory investigations: Complete blood picture , kidney function tests, liver function tests ,prothrombin time and concentration
  3. Abdominal Ultrasound
  4. Ascitic fluid paracentesis will be done to test for total leucocyte count and polymorphonuclear count , total protein and albumin levels. Testing for cytological analysis and culture will be done.
  Interventions: Procedure: paracentesis

INTERVENTIONS:
Procedure: paracentesis — paracentesis will be done for all patient for ascitic fluid study and ascitic fluid culture

SUMMARY:
Spontaneous bacterial peritonitis is defined as the presence of an infection in a previously sterile ascites in the absence of an intra-abdominal source of infection or malignancy .

The variants of Spontaneous bacterial peritonitis includes - (i) Classic Spontaneous bacterial peritonitis: -ascitic fluid polymorphonuclear leukocyte counts more than 250/mm3 and positive culture. (ii) Culture negative neutrocytic ascitis but the ascitic fluid polymorphonuclear leukocyte counts more than 250/mm3 and (iii) Bacterascites: - a culture positive ascitic fluid but the polymorphonuclear leukocyte counts less than 250/mm3

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis is a serious complication in patient with decompensated liver cirrhosis . The incidence in ascetic patients varies between 7-30 % as a consequence result of impaired defense mechanism and increased susceptibility to bacterial infection in cirrhotic patients with ascites Spontaneous bacterial peritonitis may complicated by hepatorenal syndrome or systemic sepsis and has high recurrence rate - estimated as approximately 70% within 1 year of follow up .

The clinical detection of spontaneous bacterial peritonitis requires a high index of suspicion because symptoms and signs of infection are obscure in most of patients.

About 13% of patients are asymptomatic and a few studies reported the incidence of asymptomatic spontaneous bacterial peritonitis in cirrhotic patients with ascites The most common clinical manifestations defined by Jeffries et al and Castellote et al in 2007 are: temperature above 38 °C or below 36.5 °C, chills, abdominal tenderness suggestive of peritonitis, developing or worsening hepatic encephalopathy, acute renal failure (defined by an increase in the serum creatinine level to above 133 μmol/L) and arterial hypotension (systolic arterial pressure below 80 mmHg).

The American Association for the Study of Liver Diseases recommends performing exploratory paracentesis in each patient with cirrhosis and ascites .

A study was done in Poland in 2011, shows the prevalence of spontaneous bacterial peritonitis in asymptomatic inpatients with decompensated liver cirrhosis and found that two of 37 asymptomatic cirrhotics who were included in the study met criteria of asymptomatic spontaneous bacterial peritonitis (5%) .

A french study was done in 2013 in asymptomatic cirrhotic outpatients and found that the incidence of asymptomatic Spontaneous bacterial peritonitis was only 1.2% .

Another study was done in Pakistan in 2015 and found that the incidence of asymptomatic spontaneous bacterial peritonitis in outpatient patient with cirrhosis was 10%(8 out of 80).

Another Egyptian study was done in 2016 on asymptomatic spontaneous bacterial peritonitis in adult Egyptian patient with decompensated cirrhosis and found that 21 (13%) patient was asymptomatic spontaneous bacterial peritonitis out of 160 cirrhotic patient ascetic patient who fulfill the inclusion criteria .

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with decompensated liver cirrhosis with ascites (Child B and C) regardless of the etiology of liver cirrhosis

Exclusion Criteria:

1. Symptomatic spontaneous bacterial peritonitis (patients with fever, abdominal pain or tenderness, leucocytosis, hepatic encephalopathy, impaired renal function)
2. Patients taking antibiotics for any other infections within 2 weeks e.g. pneumonia, urinary tract infection..etc
3. Patients taking antibiotics as prophylaxis for spontaneous bacterial peritonitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with decompensated liver cirrhosis with ascites (Child B and C) admitted to to AL-RAJHI LIVER HOSPITAL in assuit university for any cause other than symptomatic bacterial peritonitis(patient with fever , abdominal pain , or tenderness, leucocytosis, hepatic encephalopathy, impaired renal function) or taking antibiotics for any other infections within 2 weeks e.g. pneumonia, urinary tract infection..etc, or Patients taking antibiotics as prophylaxis for spontaneous bacterial peritonitis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
assess the frequency of asymptomatic spontaneous bacterial peritonitis in patient with decompensated liver cirrhosis admitted to Al-Rajhi Liver Hospital | 2 days
  Number of asymptomatic spontaneous bacterial peritonitis

SECONDARY OUTCOMES:
Determine the causative organisms of asymptomatic spontaneous bacterial peritonitis.. | 2 days
  making ascitic fluid culture

OTHER OUTCOMES:
Assess the efficacy of treatment in these asymptomatic patients | 2 days
  Patients whose results will confirm spontaneous bacterial peritonitis will receive treatment in the form of Cefotaxime 2gm/12 hours and then follow up by ascitic fluid testing will be done again

CONTACTS AND LOCATIONS:
Overall Officials: Antony Georgy, MBBCh, Principal Investigator — Assiut University
Locations (1):
- Al-RAhjhy Assuit unviersity hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fernandez J, Navasa M, Planas R, Montoliu S, Monfort D, Soriano G, Vila C, Pardo A, Quintero E, Vargas V, Such J, Gines P, Arroyo V. Primary prophylaxis of spontaneous bacterial peritonitis delays hepatorenal syndrome and improves survival in cirrhosis. Gastroenterology. 2007 Sep;133(3):818-24. doi: 10.1053/j.gastro.2007.06.065. Epub 2007 Jul 3. PMID 17854593
- [Result] Koulaouzidis A, Bhat S, Saeed AA. Spontaneous bacterial peritonitis. World J Gastroenterol. 2009 Mar 7;15(9):1042-9. doi: 10.3748/wjg.15.1042. PMID 19266595
- [Result] Runyon BA; AASLD Practice Guidelines Committee. Management of adult patients with ascites due to cirrhosis: an update. Hepatology. 2009 Jun;49(6):2087-107. doi: 10.1002/hep.22853. No abstract available. PMID 19475696
- [Result] Pluta A, Gutkowski K, Hartleb M. Coagulopathy in liver diseases. Adv Med Sci. 2010;55(1):16-21. doi: 10.2478/v10039-010-0018-3. PMID 20513645
- [Result] Sheer TA, Runyon BA. Spontaneous bacterial peritonitis. Dig Dis. 2005;23(1):39-46. doi: 10.1159/000084724. PMID 15920324
- [Result] Riordan SM, Williams R. The intestinal flora and bacterial infection in cirrhosis. J Hepatol. 2006 Nov;45(5):744-57. doi: 10.1016/j.jhep.2006.08.001. Epub 2006 Sep 1. No abstract available. PMID 16979776
- [Result] Nousbaum JB, Cadranel JF, Nahon P, Khac EN, Moreau R, Thevenot T, Silvain C, Bureau C, Nouel O, Pilette C, Paupard T, Vanbiervliet G, Oberti F, Davion T, Jouannaud V, Roche B, Bernard PH, Beaulieu S, Danne O, Thabut D, Chagneau-Derrode C, de Ledinghen V, Mathurin P, Pauwels A, Bronowicki JP, Habersetzer F, Abergel A, Audigier JC, Sapey T, Grange JD, Tran A; Club Francophone pour l'Etude de l'Hypertension Portale; Association Nationale des Hepato-Gastroenterologues des Hopitaux Generaux de France. Diagnostic accuracy of the Multistix 8 SG reagent strip in diagnosis of spontaneous bacterial peritonitis. Hepatology. 2007 May;45(5):1275-81. doi: 10.1002/hep.21588. PMID 17464969
- [Result] Kasztelan-Szczerbinska B, Slomka M, Celinski K, Serwacki M, Szczerbinski M, Cichoz-Lach H. Prevalence of spontaneous bacterial peritonitis in asymptomatic inpatients with decompensated liver cirrhosis - a pilot study. Adv Med Sci. 2011;56(1):13-7. doi: 10.2478/v10039-011-0010-6. PMID 21536540
- [Result] Cadranel JF, Nousbaum JB, Bessaguet C, Nahon P, Nguyen-Khac E, Moreau R, Thevenot T, Silvain C, Bureau C, Nouel O, Pilette C, Paupard T, Pauwels A, Sapey T, Grange JD, Tran A. Low incidence of spontaneous bacterial peritonitis in asymptomatic cirrhotic outpatients. World J Hepatol. 2013 Mar 27;5(3):104-8. doi: 10.4254/wjh.v5.i3.104. PMID 23556041